CLINICAL TRIAL: NCT05891548
Title: ODYSSEY: A Phase 2b Study of Suprachoroidally Administered CLS-AX in Participants With Neovascular Age-Related Macular Degeneration
Brief Title: Study to Evaluate Suprachoroidally Administered CLS-AX in the Treatment of Neovascular Age-Related Macular Degeneration
Acronym: ODYSSEY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS1002-202
Record Dates: First submitted 2023-05-24; First posted 2023-06-07 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; Wet AMD; Suprachoroidal; Tyrosine kinase inhibitor; Microinjector; Suprachoroidal Space (SCS)
MeSH Terms: conditions — Choroidal Effusions | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two treatment groups in parallel for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, Sponsor, Principal (non-injecting) Investigator, medical monitor, study coordinator, visual acuity technician, photographer, central reading center, and central laboratory will be masked to treatment assignment for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1.0 mg CLS-AX (Experimental): Suprachoroidal injection of 10 mg/mL (1.0 mg in 0.1 mL) of CLS-AX
  Interventions: Drug: CLS-AX
- Aflibercept (Active Comparator): Intravitreal injection of aflibercept (2 mg in 0.05 mL)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: CLS-AX — CLS-AX will be administered by suprachoroidal injection into the study eye on Day 1 and then every 12 to 24 weeks as determined by protocol-defined disease activity criteria.
  Other Names: axitinib injectable suspension
  Arms: 1.0 mg CLS-AX
Drug: Aflibercept — Aflibercept will be administered by intravitreal injection into the study eye once every 8 weeks (Q8W).
  Other Names: Eylea
  Arms: Aflibercept

SUMMARY:
Phase 2b, randomized, double-masked, parallel-group, active-controlled, multicenter, 36-week study designed to assess the safety and efficacy of suprachoroidally administered CLS-AX 1.0 mg with a flexible dosing regimen in participants with neovascular age-related macular degeneration previously treated with intravitreal anti-vascular endothelial growth factor (VEGF) standard of care therapy. Only one eye will be chosen as the study eye.

DETAILED DESCRIPTION:
Phase 2b, randomized, double-masked, parallel-group, active-controlled, multicenter, 36-week study designed to assess the safety and efficacy of suprachoroidally administered CLS-AX 1.0 mg with a flexible dosing regimen in participants with neovascular age-related macular degeneration previously treated with intravitreal anti-VEGF standard of care therapy. Active-control will be 2 mg intravitreal injections of aflibercept dosed per the EYLEA Prescribing Information. Only one eye will be chosen as the study eye.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration (nAMD) in the study eye within 36 months of Visit 1.
* Subfoveal choroidal neovascularization (CNV) secondary to nAMD of any lesion type in the study eye that shows total lesion area ≤30 mm2, CNV component area of ≥50% of the total lesion area, and and CNV must not be associated with subfoveal hemorrhage, subfoveal fibrosis, or subfoveal atrophy.
* Previous treatment in the study eye with between 2 and 4 anti-VEGF intravitreal injections for nAMD (faricimab, ranibizumab, bevacizumab, brolucizumab, or aflibercept) per standard of care within 6 months of Visit 1.
* History of response to prior intravitreal anti-VEGF treatment in the study eye.
* ETDRS BCVA of between 20 and 80 letters (inclusive) in the study eye.

Key Exclusion Criteria:

* ETDRS BCVA <20 letters in the study eye.
* Central subfield thickness > 400 μm or retinal pigment epithelium detachment thickness >400 μm on SD-OCT in the study eye.
* Subretinal hemorrhage, fibrosis or atrophy of >50% of the total lesion area and/or that involves the fovea on fundus fluorescein angiography and/or color fundus photography in the study eye.
* CNV due to causes other than AMD, such are ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis, in the study eye.
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Evaluations of Outcomes Related to ETDRS BCVA in the Study Eye Over Time | Baseline, Weeks 4, 12, 16, 20, 24, 28, 32 and 36
  Best Corrected Visual Acuity (BCVA) letter score measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at a starting test distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable). An increase in BCVA letter score from baseline indicates an improvement in visual acuity.

SECONDARY OUTCOMES:
Evaluations of Outcomes Related to Fluid Detected on Optical Coherence Tomography in the Study Eye Over Time | Baseline, Weeks 4, 12, 16, 20, 24, 28, 32 and 36
  Spectral-domain optical coherence tomography (SD-OCT) is a non-invasive diagnostic technique that provides high-resolution, cross-sectional tissue imaging and analysis of structural changes in the eye during disease progression. A central reading center will provide measurements and standardized gradings of outcomes related to retinal thickness and fluid in the eye, respectively.
  Central subfield retinal thickness (CST) is defined as the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE) in millimeters in the circular region centered on the anatomic fovea with a radius of 500 microns.
  The presence and location of intraretinal and subretinal fluid in the central subfield (center 1 mm) is graded as Absent (the best grade attainable); Definite, outside center subfield; Definite, center subfield involved; and Definite, both center subfield and outer subfields involved.
Evaluations of Outcomes Related to Lesion Size on Fundus Fluorescein Angiography in the Study Eye Over Time | Baseline, Week 36
  Fundus fluorescein angiography (FFA) is an invasive diagnostic procedure used to assess the anatomy, physiology, and pathology of retinal and choroidal circulation. It involves injecting fluorescein dye into a vein in the arm/hand and taking pictures as it circulates through the eye. A central reading center will provide measurements of outcomes related to the size of lesions/leakage in the eye.
  Total area of Choroidal Neovascularization (CNV) includes classic and occult components and ranges from 0-42 mm2, with 0 mm2 being the best measurement attainable.
  Total lesion area includes the total CNV and associated lesion components and ranges from 0-42 mm2, with 0 mm2 being the best measurement attainable.
  Total area of leakage includes the total area leakage from neovascularization and ranges from 0-42 mm2, with 0 mm2 being the best measurement attainable.
Evaluation of the Number of Study Drug Injections and Supplemental Therapy Injections in the Study Eye Over Time | From Baseline Through Week 36
  Number of masked study drug injections and supplemental therapy injections administered in the study eye.
Evaluation of Serious Adverse Events (SAEs) and Treatment-Emergent Adverse Events (TEAEs) | From first dose of masked study drug through the end of the study (up to 36 weeks)
  The analysis of serious adverse events (SAEs) includes both ocular and non-ocular (systemic) adverse events (AEs) meeting SAE criteria as defined in International Conference on Harmonisation (ICH) E6 Good Clinical Practice Consolidated Guidance. TEAEs are defined as adverse events that emerge during or after treatment with masked treatment having been absent pre-treatment or worsens relative to the pre-treatment state.
  Investigators will seek information on AEs at each contact with the participant. All AEs are recorded and the Investigator will independently assess seriousness, severity, and causality of each AE.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Coultas, PhD, Study Director — Clearside Biomedical, Inc.
Locations (32):
- United States (32):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Consultants of Orange County, Fullerton, California
  - Northern California Retina Vitreous Associates Medical Group, Inc, Mountain View, California
  - Retina Consultants San Diego, Poway, California
  - Retinal Consultants of Southern California, Redlands, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina, PC, Marietta, Georgia
  - Illinois Retina Associates, Oak Park, Illinois
  - Wolfe Eye Clinic, Des Moines, Iowa
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular LLC, Bloomfield, New Jersey
  - Western Carolina Retinal Associates P.A., Asheville, North Carolina
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates - Arlington, Arlington, Texas
  - Austin Retina, Austin, Texas
  - Retina Consultants of Texas-Bellairre, Bellaire, Texas
  - Texas Retina Associates - Dallas, Dallas, Texas
  - Retina Consultants of Texas - Katy, Katy, Texas
  - Texas Retina Associates-Plano, Plano, Texas
  - Retina Consultants of Texas-San Antonio, San Antonio, Texas
  - Retina Group of Washington, Fairfax, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No